CLINICAL TRIAL: NCT03649776
Title: Training Community Members in Mental Health First Aid
Brief Title: Training Church Leaders in Mental Health First Aid
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Sidney Hankerson, MD, MBA, Research Scientist, Research Foundation for Mental Hygiene, Inc.
Other Study IDs: 7224
Record Dates: First submitted 2018-07-13; First posted 2018-08-28 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Stigma
Keywords: Disparities
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mental Health First Aid — Mental Health First Aid (MHFA) is listed in the Substance Abuse and Mental Health Services Administration's National Registry of Evidence-based Programs and Practices. The program also teaches the common risk factors and warning signs of specific types of illnesses like anxiety, depression, substance use, bipolar disorder, eating disorders, and schizophrenia. Participants are introduced to local mental health resources, national organizations, support groups, and online tools for mental health and addictions treatment and support.

SUMMARY:
The purpose of this study is to train Church Leaders and other community members in Mental Health First Aid (MHFA), which is an evidence-based public mental health education program. MHFA has been found to improve people's recognition of emotional and mental health challenges and to increase people's confidence in providing help to others. Information about MHFA can be accessed at http://www.mentalhealthfirstaid.org.

MHFA consists an 8-hour training program in which participants will be provided a manual, learn the signs and symptoms of common mental health problems, and learn a 5-step action plan to help someone in an emotional crisis.

Participants ware recruited from faith-based organizations (i.e., churches), health care organizations (i.e., hospitals), and other community based organizations. There will be no treatment directly provided as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Able to provide signed formed consent

Exclusion Criteria:

* Any circumstances limiting participant's ability to complete the 8-hour training
* Inability to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This protocol primarily targets African Americans who live in Central Harlem, New York.
  Community members will also include church leaders and lay participants from local churches, health care organizations, and other community-based organizations. This will include any adult who meets study eligibility criteria and consents to take the MHFA training at one of our approved study sites. Examples of community study sites are First Corinthian Baptist Church, New York State Psychiatric Institute, and the Columbia University Wellness Center
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2016-02-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Confidence in Providing Help at 3 months | 3 months
  After reading a clinical vignette that describes a person with either Schizophrenia or Major Depression, participants are asked "How confident do you feel in helping this person?"
  Possible responses are on a 5-point Likert scale with 1 = Not at all confident and 5 = Extremely confident

SECONDARY OUTCOMES:
Change from Baseline in Stigma at 3 months | 3 months
  Personal and Perceived Stigma Scale. It is a 14-item measure that assesses stigmatizing attitudes. Questions are on a 5-point Likert scale with 1 = Strongly Agree and 5 = Strongly Disagree with scores ranging from 14 to 70. A higher score indicates greater stigma
  A clinical vignette, describing either a case with Schizophrenia or Major Depression, is presented. Participants are asked questions about social stigma, which assesses what participants' perceptions of people in their community, and personal stigma, which assesses the participants' personal beliefs.
Change from Baseline in Functional Health Status at 3 months | 3 months
  The Medical Outcomes Study 12-Item Short Form Survey Instrument (SF-12) is a validated functional health status assessment that assesses health status over the preceding 4 weeks. Measures include
  1. General Health: 5-point Likert scale with 1 = Excellent and 5 = Poor
  2. Physical Functioning: 3-point Likert scale with 1 = Yes, Limited a lot and 3 = No, Not Limited at all
  3. Role limitations resulting from physical health problems: Possible responses are 'Yes' or 'No'
  4. Role limitations resulting from emotional problems: Possible responses are 'Yes' or 'No'
  5. Bodily Pain: 5-point Likert scale with 1 = Not at All and 5 = Extremely
  6. Vitality (energy and fatigue):
  7. Mental Health: 6-point Likert scale with 1 = All of the Time and 6 = None of the Time
  8. Social Functioning: 6-point Likert scale with 1 = All of the Time and 6 = None of the Time Total Scores range from 0 to 100, with higher scores indicating poorer health

OTHER OUTCOMES:
Semi structured Interviews at 3 months | 3 months
  Semi-structured interviews are conducted with participants either over the telephone, in-person at their church or at the New York State Psychiatric Institute. The purpose of the interview is to get examples of how participants utilized the skills in Mental Health First Aid training, what action items they completed, and how the training could be improved for use among other communities

CONTACTS AND LOCATIONS:
Overall Officials: Sidney H Hankerson, MD, MBA, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Describes the Mental Health First Aid intervention — https://www.mentalhealthfirstaid.org/
- See also: Describes the Community Advisory Board created by Dr. Hankerson's NIMH-funded K23 Career Development Award. This Community Advisory Board selected Mental Health First Aid as the study intervention. — https://www.communitycoalitionformentalhealth.com/

DOCUMENTS (1):
  • Study Protocol (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT03649776/Prot_000.pdf